CLINICAL TRIAL: NCT05950750
Title: Turkey Thrombotic Thrombocytopenic Purpura Disease Registry: National Multicenter Study
Status: Recruiting | Type: Observational
Sponsor: Turkish Hematology Association (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: eTTP-THD
Record Dates: First submitted 2023-01-31; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: TTP - Thrombotic Thrombocytopenic Purpura
Keywords: TTP; THD
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Patients: Non interventional observational

SUMMARY:
21 hematology centers in Turkey will participate in this noninterventional observational study. The recruitment target is 960 cases. Patients will be followed-up at least 1 year or to the end of the study according to the physicians' discretion, or withdrawal of consent. Recruitment period will be 36 months. Data will be collected via electronic case report form. Since the study cohort does not include only newly diagnosed patients, all aTTP patients will be included to the study, previous treatments and diagnosis information data could also be collected from hospital records. Patients recruitment duration: 3 years (36 months) Patients follow-up duration: 1 year (12 months)

DETAILED DESCRIPTION:
Because of the non-interventional nature of the study, there is no predefined treatment protocol. The patients will be treated according to the routine practices of the centers. In observational drug studies, the drug to be administered in treatment should be prescribed and patient's treatment should be started prior to study inclusion decision is made as a principle. The participating physician will continue to treat the patients according to their routine practices. Not only newly diagnosed patients, all aTTP patients within participated centers will be recruited and 12 months follow-up data will be collected. 21 hematology centers in Turkey will participate in this noninterventional observational study. The recruitment target is 960 cases. Patients will be followed-up at least 1 year or to the end of the study according to the physicians' discretion, or withdrawal of consent. Recruitment period will be 36 months. Data will be collected via electronic case report form. Since the study cohort does not include only newly diagnosed patients, all aTTP patients will be included to the study, previous treatments and diagnosis information data could also be collected from hospital records. Patients recruitment duration: 3 years (36 months) Patients follow-up duration: 1 year (12 months)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as aTTP after 01.01.2015
* Patients with ADAMS13<10%
* Thrombocytopenia (<100.000)
* Coombs (-)
* Microangiopathic hemolytic amenia
* 18 years and older

Exclusion Criteria:

- Patient who does not sign informed consent form

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with TTP and signed an informed written consent will be included into the study. Because of the non-interventional nature of the study, there is no predefined treatment protocol. The patients will be treated according to the routine practices of the centers. In observational drug studies, the drug to be administered in treatment should be prescribed and patient's treatment should be started prior to study inclusion decision is made as a principle. The participating physician will continue to treat the patients according to their routine practices. Not only newly diagnosed patients, all aTTP patients within participated centers will be recruited and 12 months follow-up data will be collected.
Sampling Method: Probability Sample
Enrollment: 960 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-12-21 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Number of episodes | Through study completion, an average of 4 years
  Median number of episodes will be given
To describe treatment patterns among TTP patients | Through study completion, an average of 4 years
  All treatments received by patients will be expressed as percentages

SECONDARY OUTCOMES:
To describe demographic characteristics of TTP patients | 24 months
  Age, sex, family history, comorbidities will be expressed as percentages

CONTACTS AND LOCATIONS:
Overall Officials: ilker kurkcu, Study Director — Sentez-CRO
Locations (1):
- Baskent Universtiy Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karakus S, Bakanay SM, Kalayoglu Besisik S, Eskazan AE, Ayyildiz O, Gurkan E, Salim O, Karakus V, Guler N, Keklik M, Ozcebe OI, Ozkalemkas F, Ozkocaman V, Yilmaz U, Dadin S, Ucar MA, Sonmez M, Karakus A, Atas U, Koc LZ, Gunduz E, Kabukcu Hacioglu S, Unver Koluman B, Ozet G, Guney T, Fidan K, Karaagac Akyol T, Kikili CI, Demirkan F, Yavasoglu I, Dagtas S, Kestane M, Uskudar Teke H, Kocak Toprak S, Karatas A, Yagci M, Ozatli D, Ozkurt ZN, Ilhan O, Ar MC. Clinical Manifestations, Treatment Characteristics, and Clinical Outcomes in Patients with Immune Thrombotic Thrombocytopenic Purpura (iTTP) in a Real-World Setting: An Interim Analysis of the Turkish iTTP Registry. Turk J Haematol. 2025 Aug 29;42(3):203-212. doi: 10.4274/tjh.galenos.2025.2025.0134. Epub 2025 Jul 23. PMID 40699136